CLINICAL TRIAL: NCT03408184
Title: Comparison Between Lumbar Paravertebral and Field Blocks in Pediatric Inguinal Hernia Surgery.
Brief Title: Lumbar Paravertebral in Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MS/16.06.19
Record Dates: First submitted 2018-01-10; First posted 2018-01-23 (Actual); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar paravertebral group (Active Comparator): After general anesthesia, the patient is placed prone. To establish the level of the block, we used US-counting of vertebrae. After determining the lumbar one level, the block performed at a parallel line 2 cm lateral to the spinous process, the transducer is moved until the corresponding transverse process is identified. Utilizing an in-plane approach from lateral to medial, a spinal needle is advanced until contact with the transverse process. The needle is withdrawn and redirected caudally under the transverse process helped by the loss of resistance technique. the solution is slowly injected after negative aspiration for blood.
  Interventions: Drug: Lumbar paravertebral group
- The field block group (Active Comparator): The ilioinguinal nerve block was done at one fingerbreadth from the anterior superior iliac spine in a line with the pubic tubercle, The injection was done after the bob of the needle after passing the external oblique aponeurosis and muscle and 5ml of the solution is injected. The rest of the solution is injected in the incision line.
  Interventions: Drug: The field block group

INTERVENTIONS:
Drug: Lumbar paravertebral group — A mixture of 0.5 ml /kg bupivacaine (0.25%), and 0.5µg/Kg dexmedetomidine and Epinephrine 5 microgram/ ml.
  Arms: Lumbar paravertebral group
Drug: The field block group — A mixture of 0.5 ml /kg bupivacaine (0.25%), and 0.5µg/Kg dexmedetomidine and Epinephrine 5 microgram/ ml.
  Arms: The field block group

SUMMARY:
An inguinal hernia is one of the most common disorders requiring surgical repair in pediatrics. The effective treatment of postoperative pain in infants and children is challenging. Although the use of opioid analgesics is generally safe, adverse effects occur frequently, so the use of alternative analgesic techniques when available to improve postoperative analgesia while limiting opioid-related adverse effects, that is why there is an increase in the use of regional anesthetic techniques in infants and children.

DETAILED DESCRIPTION:
Different anesthetic regional techniques can be used for anesthesia and analgesia of the lower abdominal surgeries such as caudal, spinal, epidural, transversus abdominis plane block, ilioinguinal nerve block, lumbar plexus block, the field block and abdominal paravertebral block. The use of regional anesthesia with ultrasound guidance can help decrease complications of regional blocks.

In the lumbar area, the lumbar paravertebral space is a potential space formed by the vertebral bodies, intervertebral discs and intervertebral foramina medially, the psoas major muscle anterolaterally and the erector spinae muscles, the transverse process and intertransverse ligaments posteriorly. There is no costotransverse ligament in the lumbar region. The lumbar spinal nerve roots run through the paravertebral space then continue through the psoas major muscle where they form the lumbar plexus.The spinal nerves in this space are devoid of a fascial sheath making them exceptionally susceptible to local anesthetics. The diaphragm and psoas muscle separate the thoracic and lumbar paravertebral areas; however, communication may occur via the medial and lateral arcuate ligaments of the diaphragm.

Field block can be done by subcutaneous injection of a local anesthetic in an area bordering on the field to be anesthetized. It is safe, simple, effective, and economical, without post anesthesia side effects. Furthermore, local anesthesia administered before the incision produces longer postoperative analgesia because of local infiltration, theoretically, inhibits the build-up of local nociceptive molecules, and therefore, there is better pain control in the postoperative period.

The aim of this study is to compare the analgesic and autonomic effects of unilateral abdominal ultrasound guided paravertebral block with field block in pediatric inguinal hernia surgery.

This study hypothesizes that unilateral abdominal ultrasound guided paravertebral block may be more superior to field block in reducing intra and postoperative pain in the pediatric inguinal hernia. The analgesic efficacy and duration of ultrasound (US) guided unilateral lumbar paravertebral block and field block were compared when dexmedetomidine and epinephrine were added as adjuvants to bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

1. Patients subjected to an elective unilateral inguinal hernia repair.
2. American Society for Anesthesiologists physical status grades I and II.

Exclusion Criteria:

1. Parental refusal. 2. Neuromuscular diseases (as myopathies, myasthenia gravies, etc.) 3. Hematological diseases, bleeding or coagulation abnormality. 4. Psychiatric diseases. 5. Local skin infection and sepsis at the site of the block. 6. Known intolerance to the study drugs.

-

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
The total dose of analgesics required in the post-operative periods | 24 hours postoperatively
  Fentanyl in microgram.

SECONDARY OUTCOMES:
Modified Faces Legs Activity Cry Consolability Revised pain Scale | postoperative at 1, 2, 4, 8,16, 24 hours.
  pain score of 5 items (Faces, Legs, Activity, Cry, Consolability) each of 0, 1, or 2 points. 0= express no pain, 1= mild pain, 2= the highest pain indicator. A total score 0 = Relaxed and comfortable. 1-3 = Mild discomfort. 4-6 = Moderate pain. 7-10 = Severe pain.
Mean Blood pressure | Basal preoperative, during incision, 30 minutes, 60 minutes intraoperatively, postoperative at 1, 2, 4, 8,16, 24 hours.
  millimeter mercury
Heart rate | Basal preoperative, during incision, 30 minutes, 60 minutes intraoperatively, postoperative at 1, 2, 4, 8,16, 24 hours.
  beat/minutes
Modified Ramsay sedation scale. | postoperative at 2, 4, 6, 12, 16, 24 hours.
  a scale from (1- 6), 1 = anxious; 2 = oriented & tranquil; 3 = sedated, but responds to commands; 4 = asleep, brisk glabellar reflex or response to loud noise; 5 = asleep, slugglish glabellar reflex or response to loud noise; 6 = asleep with no response to painful stimulus
Parents' satisfaction score | postoperative after 24 hours.
  in a visual analogue score from (0-10), 0= minimal satisfaction, 10 = the highest satisfaction.
Adverse effects including nausea and vomiting, bradycardia (heart rate less than 60 beat/minute) | postoperatively in the first 24 hours.
  percent

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Children's Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
after publication
Supporting Information: SAP, CSR
Time Frame: no limit
Access Criteria: e mail: ayatebrahimeid@gmail.com